CLINICAL TRIAL: NCT06890572
Title: Clinical Validation of the Efficacy of Air Purifiers Equipped With Harmful Gas Filters in Improving Indoor Environment and Alleviating Allergic Symptoms in Allergic Rhinitis Patients
Brief Title: Validation of the Efficacy of Air Purifiers in Indoor Environment and Allergic Symptoms in Allergic Rhinitis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: LG Electronics Inc. (Industry)
Responsible Party: Principal Investigator, Park Kyung Hee, Clinical Associate Professor, Yonsei University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2024-1043
Record Dates: First submitted 2025-02-26; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Rhinitis Allergic
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre-placebo/post-Intervention group (Other): Group A will receive a fake air purifier during study period 1, and during study 2, the HEPA+VOC filter air purifier will be operated.
  Interventions: Device: HEPA + VOC collecting filter purifier; Device: fake air purifier
- pre-Intervention/post-placebo group (Other): Group A will receive the HEPA+VOC filter air purifier during study period 1, and during study 2, a fake air purifier will be operated.
  Interventions: Device: HEPA + VOC collecting filter purifier; Device: fake air purifier

INTERVENTIONS:
Device: HEPA + VOC collecting filter purifier — Subjects operate HEPA + VOC collecting filter purifier
Device: fake air purifier — Subjects operate fake air purifiers

SUMMARY:
This study targets adult patients between the ages of 19 and 60 who were diagnosed with allergic rhinitis caused by indoor inhalation antigens. Patients with moderate to severe and persistent allergic rhinitis who continue to require medication such as antihistamines and nasal spray steroids for allergic rhinitis are the subjects of this study.

Patients who participate in the study will install air purifiers for a certain period of time and observe the objective and subjective improvement of rhinitis symptoms. The study is conducted on two separate occasions for four weeks, and there is a two-week period between the two periods of no use of air purifiers. There are two types of air purifiers:

1)It is an air purifier with a HEPA filter and a VOC filter, and 2) a fake air purifier without air cleaning function.

Subjects are divided into Group A and Group B. Group A will receive a fake air purifier, and Group B will be assigned an air purifier with a HEPA + VOC collecting filter. After using the assigned air purifier for the first four weeks, you will have a period of not using it for two weeks, and then replace the air purifiers with each other and use it again for four weeks. When you first assign an air purifier, you will receive an air purifier with a certain filter It is randomly assigned without knowing whether both the researcher and the patient will receive a regular period.

During the study period, patients need to visit three times, including when registering for the study, and the study period is screened It will take about 5 months from the end of the air purifier operation

DETAILED DESCRIPTION:
This study targets adult patients between the ages of 19 and 60 who were diagnosed with allergic rhinitis caused by indoor inhalation antigens. Patients with moderate to severe and persistent allergic rhinitis who continue to require medication such as antihistamines and nasal spray steroids for allergic rhinitis are the subjects of this study.

Patients who participate in the study will install air purifiers for a certain period of time and observe the objective and subjective improvement of rhinitis symptoms. The study is conducted on two separate occasions for four weeks, and there is a two-week period between the two periods of no use of air purifiers. There are two types of air purifiers:

1)It is an air purifier with a HEPA filter and a VOC filter, and 2) a fake air purifier without air cleaning function.

Subjects are divided into Group A and Group B. Group A will receive a fake air purifier, and Group B will be assigned an air purifier with a HEPA + VOC collecting filter. After using the assigned air purifier for the first four weeks, you will have a period of not using it for two weeks, and then replace the air purifiers with each other and use it again for four weeks. When you first assign an air purifier, you will receive an air purifier with a certain filter It is randomly assigned without knowing whether both the researcher and the patient will receive a regular period.

During the study period, patients need to visit three times, including when registering for the study, and the study period is screened It will take about 5 months from the end of the air purifier operation

A detailed chronological overview of the study is as follows

1. Screening and Baseline Visits (Visit 1) Before the process of the study begins, the study subjects are fully explained about the entire research process and checked whether they meet the selection and exclusion criteria. If the selection criteria are met, a written consent form will be written, basic demographic information (gender, age, medical history (including allergic disease-related and surgical history), and drug administration history (four weeks before registration). We will conduct a survey on subjective symptoms of allergic rhinitis, drug use scores, subjective score indicators, and quality of life evaluation indicators, and double-check the drugs currently being taken by the study subjects.

   If you have previously used drugs for allergic rhinitis, you can maintain the medication without change and prescribe additional relief drugs if necessary.
2. Installation of air purifier and Study I after randomization Randomization is a method that is divided into groups A and B and is assigned based on a randomized list (random table) with statistician advice at a ratio of 1:1 respectively.

   The first study (Study I) will run for four weeks. During this period, the air purifier will continue to operate, and no indoor ventilation will be performed for these four weeks to reduce other factors that may affect indoor air quality. After four weeks, the air purifier will be remotely controlled, and indoor air quality information will be continuously collected in the filter replacement.
3. Interim Visit (Visit 2) The subject of the study will visit the hospital with a journal written about the changes in symptoms and the use of drugs after the first operation of the purifier (Study I). During the first and second visits, the symptoms will be checked for differences and whether relief drugs have been used, and additional relief drugs will be prescribed if necessary, along with retraining on the next visit schedule.
4. Study II progress and end visit after replacement of air purifier filter (Visit 3) To proceed with the second study (Study II), LG Electronics installers revisit each home and install Dual Defense Filter (HEPA + VOC capture filter) in Group A. Conversely, Group B will remove the Dual Defense filter and attach void labels again each. Study II will also run for four weeks, during which the air purifier is continuously running and there is no indoor ventilation.

The subject of the study should visit the hospital with symptoms and drug use log even at the end of the visit, and the change in symptoms and the use of relief drugs will be confirmed. At the end of the study, we will disclose which group the study subjects were assigned to.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 19 to 60
* A person with moderate-severe persistent allergic rhinitis diagnosed by an allergy specialist or otolaryngologist and maintained without any change in treatment for more than one month
* Total nasal symptom Score ≥ 8
* Patients with allergic rhinitis caused by indoor inhalation antigen antigens (House dust mites ± If the wheal size of the pet skin test is greater than 3mm or the concentration of specific IgE measured by ImmunoCAP ≥ 0.35 kUA/L)
* A person who spends at least 8 hours/day per week in the home where the cleaner will be installed
* A person with a wi-fi installed in the home where the purifier will be installed
* A person who can read and write in Korean
* A person who fully explains the contents, decides to participate in the study according to his/her free will, and signs a written consent form approved by each agency IRB

Exclusion Criteria:

* Patients sensitized to seasonal antigens (tree, grass or weed pollen)
* Rhinitis patients caused by causes other than allergic rhinitis (drug rhinitis, vascular rhinitis, infectious rhinitis, etc.)
* Anyone who has required more than 2 weeks of systemic steroid use in the last 3 months
* A person taking antihistamines for reasons other than rhinitis (chronic urticaria, etc.)
* Those with anatomical abnormalities that cause nasal congestion, such as non-segmental curvature and non-segmental species
* A person who has a plan to move during the study period or is scheduled to leave where air purifiers are installed for at least five consecutive days (e.g., travel, business trip, etc.)
* A person who has already used an air purifier within the last three months
* Pregnant women, lactating women, persons lacking decision-making ability, persons accommodated in facilities
* A person whose researcher is deemed unfit to participate in clinical research due to other reasons

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-05-23 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Change of indoor total volatile organic compound concentration | up to 12 weeks
  The indoor air collected through the air purifier is analyzed to evaluate the total indoor volatile organic compound concentration.

SECONDARY OUTCOMES:
Change of indoor formaldehyde concentrations | up to 12 weeks
  Measure the indoor formaldehyde concentration through the air purifier
Change of indoor NO2 concentrations | up to 12 weeks
  Measure the indoor NO2 concentration through the air purifier
Change of indoor PM10 concentrations | up to 12 weeks
  Measure the indoor PM10 concentration through the air purifier
Change of indoor PM2.5 concentrations | up to 12 weeks
  Measure the indoor PM2.5 concentration through the air purifier
Change of indoor PM1.0 concentrations | up to 12 weeks
  Measure the indoor PM1.0 concentration through the air purifier
Change of Allergic rhinitis symptom score (Total natal symtom score) | up to 12 weeks
  TNSS has a total score of 12, and evaluate the degree of runny nose, sneezing, stuffy nose, and itchy nose. A score of 0 is no symptom, a score of 1 is mild (symptomatic/symptomatic but mild and easily tolerable), a score of 2 is moderate (symptomatic/symptomatic but tolerable), and a score of 3 is severe (symptomatic/symptomatic and difficult to bear and interfere with daily life or sleep). the higher the score, the more severe the rhinitis symptoms
Changes in the use of anti-allergic rhinitis medication (Rescue Medication Score) | up to 12 weeks
  Rescue Medication Score is evaluated from 0 to 2. A score of 0 means no additional medication, a score of 1 means additional use of oral or nasal antihistamines, and a score of 2 means additional use of nasal steroids, and a higher score means more rhinitis symptoms
A change in Quality of Life by Allergic Rhinitis | up to 12 weeks
  Evaluate using the quality of life questionnaire. The quality of life evaluation questionnaire is a questionnaire investigating the impact of allergic rhinitis on patients' lives for a week. The higher the score, with a total score of 60, the more severe the symptoms of rhinitis.
Change of odor score | up to 12 weeks
  valuate the subjective level of smell that a subject feels in the home. A score of 0 is odorless (relatively odorless and usually unable to detect anything with his or her sense of smell), a score of 1 is a sensed smell (the smell is unknown but capable of feeling the smell), a score of 2 is a normal smell (the smell is strong enough to know what it is), a score of 3 is a strong smell (the smell is strong enough to detect easily), a score of 4 is an extreme smell (a strong smell, for example, from a conventional toilet in summer), and a score of 5 is an unbearable smell (the strong smell that is difficult to endure and feels like stopping breathing). A total of five points means that the higher the score, the more severe the smell is.
Change in the time required for indoor pollutants to decrease from maximum concentration to baseline | up to 12 weeks
  Through the data collected by the air purifier, the time required for the indoor pollutant source to be reduced from the maximum concentration to the baseline is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Hee Park, Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (1):
- Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No